CLINICAL TRIAL: NCT04669366
Title: Treatment Patterns With Targeted Therapies in Metastatic Renal Cell Carcinoma (mRCC) in Sweden - A Retrospective Analysis of Data From National Registries
Brief Title: Treatment Patterns With Targeted Therapies In Mrcc In Sweden - A Retrospective Analysis Of Data From National Registries
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181234; RENCOMP3 (Other: Alias Study Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-06

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Sunitinib; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients in Sweden with metastatic renal cell carcinoma: The cohort of patients with metastatic renal cell carcinoma in Sweden
  Interventions: Drug: sunitinib; Drug: axitinib

INTERVENTIONS:
Drug: sunitinib — As provided in real world
  Other Names: Sutent
Drug: axitinib — As provided in real world
  Other Names: Inlyta

SUMMARY:
The objectives of this study is to investigate treatment patterns and outcomes for Sutent and Inlyta in mRCC patients in a nationwide population-based setting in Sweden.

ELIGIBILITY:
Inclusion Criteria:

1. all patients aged ≥ 18 years with at least one filled prescription of an oral targeted therapy relevant for treating mRCC registered in the Swedish Prescribed Drug Register (PDR) between July 1st 2005 and June 30th 2020. The Anatomical Therapeutic Chemical (ATC) codes for the oral drugs relevant for treating mRCC are the following: L01XE04 (sunitinib), L01XE05 (sorafenib), L01XE11 (pazopanib), L01XE17 (axitinib), L01XE10 (everolimus), L01XE26 (cabozantinib), L01XE34 (tivozantib), L01XE29 (lenvatinib).
2. The patients identified in the PDR that also are identified in the SCR with the International Classification of Diseases and Related Health Problems (ICD)-7 diagnosis codes I800 or I809 and ICD-10 codes C64.0 and C64.9 from January 1st 2000 until December 31st 2019;excluding ICD-7 code I801 (cancer of the renal pelvis) will be included in the analysis set.

Exclusion Criteria:

Patients with ICD-7 code I801 will be excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data used for the analyses includes all patients aged ≥ 18 years with at least one filled prescription of an oral targeted therapy relevant for treating mRCC registered in the Swedish Prescribed Drug Register between July 1st 2005 (there is no data available in the register before this date) and June 30th 2020. The Anatomical Therapeutic Chemical (ATC) codes for the oral drugs relevant for treating mRCC are the following: L01XE04 (sunitinib), L01XE05 (sorafenib), L01XE11 (pazopanib), L01XE17 (axitinib), L01XE10 (everolimus), L01XE26 (cabozantinib), L01XE34 (tivozantib), L01XE29 (lenvatinib). The patients identified in the PDR that also are identified in the SCR with the International Classification of Diseases and Related Health Problems (ICD)-7 diagnosis codes I800 or I809 and ICD-10 codes C64.0 and C64.9 from January 1st 2000 until December 31st 2019;excluding ICD-7 code I801 (cancer of the renal pelvis) will be included in the analysis set.
Sampling Method: Non-Probability Sample
Enrollment: 1205 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Innovations AB, Sollentuna, Sweden

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Jakobsson M, Strambi A, Nilsson F, Arpegard J, Dalen J. Real-world experience of second-line axitinib in metastatic renal cell carcinoma: analysis of the Swedish population. Future Oncol. 2024;20(20):1385-1392. doi: 10.1080/14796694.2024.2351352. Epub 2024 Jul 26. PMID 39057291
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with metastatic renal cell carcinoma (mRCC), aged above 18 years with at least one filled prescription of an oral targeted therapy relevant for treating mRCC, registered in the Swedish Prescribed Drug Register between 01-July-2005 and 31-Dec-2019, were included in this study and their data was observed retrospectively.
Pre-assignment Details: Participants were treated with sunitinib in the first line (1L) mRCC setting and with axitinib in the second line (2L) mRCC setting. The index date was the date of first identified prescription of the participant.
Groups:
- Sunitinib 4:2 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib on 4:2 (4 weeks on/2 weeks off) schedule in the daily clinical practice based on recommended dose in the Summary of Product Characteristics (SPC), between 01-July-2005 to 31-Dec-2019, were observed retrospectively.
- Sunitinib 2:1 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib on 2:1 (2 weeks on/1 week off) schedule in the daily clinical practice based on recommended dose in the SPC, between 01-July-2005 to 31-Dec-2019, were observed retrospectively.
- Sunitinib: Switched From 4:2 to 2:1 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib on 4:2 schedule then switched to 2:1 schedule in the daily clinical practice based on recommended dose in the SPC, between 01-July-2005 to 31-Dec-2019, were observed retrospectively.
- Axitinib: Participants with mRCC who initiated axitinib as second-line treatment in continuous 4 week cycles, between 01- July-2005 to 31-Dec-2019 based on recommended dose in the SPC, were observed retrospectively.
Period: Overall Study
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib
Started | 704 | 320 | 71 | 110
Completed | 704 | 320 | 71 | 110
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed.
Groups:
- Sunitinib 4:2 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib on 4:2 schedule in the daily clinical practice based on recommended dose in the SPC, between 01-July-2005 to 31-Dec-2019, were observed retrospectively.
- Sunitinib 2:1 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib on 2:1 schedule in the daily clinical practice based on recommended dose in the SPC, between 01-July-2005 to 31-Dec-2019, were observed retrospectively.
- Total: Total of all reporting groups
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib | Total
Number analyzed (Participants) | 704 | 320 | 71 | 110 | 1205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.58 (9.15) | 67.85 (9.70) | 66.51 (8.23) | 65.53 (9.89) | 66.82 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 103 | 25 | 26 | 363
  Male | 495 | 217 | 46 | 84 | 842
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Filled Sunitinib Prescription
Description: Number of participants who had at least one filled prescription of sunitinib were analyzed and reported in this outcome measure.
Time Frame: Data collected from index date up to 168 months (during retrospective observation period of 14 years, from 01-July-2005 to 31-Dec-2019). Index date was defined as the participant's first identified prescription date
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib
Number analyzed (Participants) | 704 | 320 | 71 | 110
Participants | 704 | 320 | 71 | 53

2. Primary Outcome: Number of Participants With 4:2 Sunitinib Schedule Without Any Modification
Description: Number of participants that initiated treatment with 4:2 (4 weeks on/2 weeks off) sunitinib schedule and did not have any modification in the schedule were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed. This outcome measure was planned to be analyzed only for Sunitinib 4:2 Schedule reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib 4:2 Schedule
Number analyzed (Participants) | 704
Participants | 704

3. Primary Outcome: Number of Participants With 2:1 Sunitinib Schedule Without Any Modification
Description: Number of participants that initiated treatment with 2:1 (2 weeks on/1 week off) sunitinib schedule and did not have any modification in the schedule were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed. This outcome measure was planned to be analyzed only for Sunitinib 2:1 Schedule reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib 2:1 Schedule
Number analyzed (Participants) | 320
Participants | 320

4. Secondary Outcome: Number of Participants Switched From 4:2 Sunitinib Schedule to 2:1 Sunitinib Schedule
Description: Number of sunitinib users that started on a 4:2 (4 weeks on/2 weeks off) schedule and later was switched to a 2:1 (2 weeks on/1 week off) schedule were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed. This outcome measure was planned to be analyzed only for Sunitinib: Switched From 4:2 to 2:1 Schedule reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4:2 to 2:1 Schedule
Number analyzed (Participants) | 71
Participants | 71

5. Secondary Outcome: Number of Participants on Second Line Treatment With at Least 1 Filled Axitinib Prescription
Description: Number of participants that had at least one filled prescription of axitinib were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed. This outcome measure was planned to be analyzed only for Axitinib reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 110
Participants | 110

6. Secondary Outcome: Time to Treatment Discontinuation (TTD)
Description: TTD was defined as the difference between the start and end-dates for a treatment episode regardless of reason for discontinuation. The start date for a treatment episode was defined as the date of first dispensed package and the end date was defined as the date of the last dispensed package with the same Anatomical Therapeutic Chemical (ATC) code, plus the number of days that package, as well as accumulated medicine was intended to cover. End date was overruled if there was a new filled prescription of another relevant ATC code or death happens before this, then either of these dates represents the end date. If no end of prescribed supply was recorded, data was censored at latest available date in data.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib
Number analyzed (Participants) | 704 | 320 | 71 | 110
Months | 4.55 [4.3 to 5.6] | 6.20 [5.6 to 7.2] | 13.91 [8.1 to 20.6] | 5.19 [3.7 to 6.1]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (number of days) from the start of the treatment (the date of the first dispensed package of Sunitinib or axitinib) until the date of death as documented in the Cause of Death Register. If no death was recorded, data was censored at latest available date in data.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from national registries and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib
Number analyzed (Participants) | 704 | 320 | 71 | 110
Months | 13.48 [12.3 to 15.8] | 21.79 [18.1 to 26.1] | 32.20 [25.1 to 48.3] | 12.23 [7.7 to 14.2]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Data collected from index date up to 168 months (during retrospective observation period of 14 years, from 01-July-2005 to 31-Dec-2019); Index date was defined as the participant's first identified prescription date
Description: Minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Arm/Group | Sunitinib 4:2 Schedule | Sunitinib 2:1 Schedule | Sunitinib: Switched From 4:2 to 2:1 Schedule | Axitinib
All-Cause Mortality (participants affected / at risk) | 627/704 | 168/320 | 53/71 | 82/110
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT04669366/Prot_SAP_000.pdf